CLINICAL TRIAL: NCT02573714
Title: Comparison of Sub-dissociative Intranasal Ketamine Plus Standard Pain Therapy Versus Standard Pain Therapy in the Treatment of Pediatric Sickle Cell Disease Vasoocclusive Crises in Resource-limited Settings: a Multi-centered, Randomized, Controlled Trial
Brief Title: Sub-dissociative Intranasal Ketamine for Pediatric Sickle Cell Pain Crises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cameroon Baptist Convention Health (Other)
Collaborators: Carolinas Medical Center (Other); Muhimbili National Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB2015-07; MNH/IRB/I/2015/14 (Other: Muhimbili National Hospital IRB); TFDA0015/CTR/0015/9 (Other: Tanzania Food and Drugs Authority); NIMR/HQ/R.8a/Vol. IX/2299 (Other: Tanzania National Institute for Medical Research)
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Sickle Cell Disease
Keywords: Ketamine; Intranasal; Pain crisis; Vasoocclusive Pain; Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Ketamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Ketamine (Experimental): Patients allocated to receive intranasal ketamine (intervention) in addition to standard pain therapy. Patients enrolled in this arm will utilize the FPS-R and follow-up PedsQL-SCD.
  Interventions: Drug: Ketamine; Other: Standard Pain Therapy; Other: Pediatric Quality of Life - Sickle Cell Disease Module; Other: Faces Pain Scale - Revised
- Normal Saline (Placebo Comparator): Patients allocated to receive intranasal normal saline (placebo) in addition to standard pain therapy. Patients enrolled in this arm will utilize the FPS-R and follow-up PedsQL-SCD.
  Interventions: Drug: Normal Saline; Other: Standard Pain Therapy; Other: Pediatric Quality of Life - Sickle Cell Disease Module; Other: Faces Pain Scale - Revised

INTERVENTIONS:
Drug: Ketamine — Intranasal ketamine (concentration: 50 mg/ml, dose: 1 mg/kg) will be given at time zero. Intranasal administration will be performed by placing the needleless syringe gently into the nares with the patient sitting upright. Volumes of ≤ 0.75ml will be nasally inhaled in a single nare, while volumes > 0.75ml will be divided between both nares. Patients who are unable to inhale the medication nasally will receive drip administration of the same volume while recumbent on the bed.
  Arms: Intranasal Ketamine
Drug: Normal Saline — Intranasal normal saline (placebo: volume-matched with intranasal ketamine) will be given at time zero. Intranasal administration will be performed by placing the needleless syringe gently into the nares with the patient sitting upright. Volumes of ≤ 0.75ml will be nasally inhaled in a single nare, while volumes > 0.75ml will be divided between both nares. Patients who are unable to inhale the medication nasally will receive drip administration of the same volume while recumbent on the bed.
  Other Names: NaCl 0.9%
  Arms: Normal Saline
Other: Standard Pain Therapy — Typical management strategy for pediatric sickle cell disease vasoocclusive crises including acetaminophen/paracetamol, ibuprofen, oral opioids, and injectable opioids depending on pain severity.
Other: Pediatric Quality of Life - Sickle Cell Disease Module — Standardized quality of life assessment performed 2-3 weeks post intranasal medication administration to evaluate pain management and severity of symptoms after discharge from the hospital.
  Other Names: PedsQL-SCD
Other: Faces Pain Scale - Revised — All patients will answer the FPS-R at 0 minutes (immediately prior to receiving intranasal medication), 30 minutes, 60 minutes, and 120 minutes to assess current pain status.
  Other Names: FPS-R

SUMMARY:
The purpose of this study is to determine if the use of ketamine, sniffed in the nose, is a safe and effective way to help reduce pain in pediatric sickle cell patients with pain crises in resource-limited settings.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, drug trial using sub-dissociative intranasal ketamine as an adjunct to standard pharmacotherapy for the management of pediatric sickle cell disease vasoocclusive pain crises in resource-poor settings. Pediatric patients will be enrolled at a teaching and referral hospital in West Africa. Patients will be randomly assigned to the treatment arm - standard therapy plus sub-dissociative intranasal ketamine (1 mg/kg) given at time zero) or the control arm - standard therapy plus intranasal normal saline (volume-matched to treatment arm), and patients will evaluated at standard intervals to assess for pain scores and vital signs (0 minutes, 30 minutes, 60 minutes, and 120 minutes). Pain will be assessed using the Faces Pain Scale - Revised (FPS-R). Patients will also be observed for any potential side effects or adverse events. All patients will be contacted 2-3 weeks post intranasal medication administration for over-the-phone follow-up using a portion of the PedsQL-SCD questionnaire, to assess for basic quality of life related to pain management and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease (SCD)
* Vasoocclusive pain crisis
* Requiring analgesia

Exclusion Criteria:

* Anatomic variations of nose precluding intranasal medication administration
* Ketamine allergy
* Non-verbal
* Obtunded
* Pregnant
* Other acute SCD complications:

  * Acute chest syndrome
  * Sepsis
  * Stroke
  * Splenic sequestration
  * Pulmonary embolism
  * Acute osteomyelitis

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline (time zero) in FPS-R scores between treatment groups | Baseline (time zero, indicated by injection of intranasal medication), 30 minutes, 60 minutes, and 120 minutes
  Measure of differences of change of FPS-R scores from baseline to 30 minutes, 60 minutes, and 120 minutes compared between treatment arms

SECONDARY OUTCOMES:
Hospital length of stay | through study completion, an average of 3 days
  Hospital length of stay recorded from time zero to time of discharge documented by the study clinician will be a secondary outcome measure.
Quality of life assessment (PedsQL-SCD Module scores) | Time of first intranasal administration to 3 weeks post intranasal intervention.
  PedsQL-SCD Module scores obtained by study clinicians using over-the-phone interviews between two-three weeks post intervention will be a secondary outcome measure.
Analgesia use - paracetamol | Time of initial intranasal drug administration to 2 hours post intranasal drug administration
  Individual evaluation of total paracetamol use per kilogram body weight
Analgesia use - ibuprofen | Time of initial intranasal drug administration to 2 hours post intranasal drug administration
  Individual evaluation of total ibuprofen use per kilogram body weight
Analgesia use - opioids | Time of initial intranasal drug administration to 2 hours post intranasal drug administration
  Individual evaluation of total opioid use expressed as morphine equivalents per body weight.

OTHER OUTCOMES:
Adverse Events | Time of initial intranasal drug administration to 2 hours post intranasal drug administration
  Adverse events include: bad taste is mouth, drowsiness, dizziness, itchy nose, nausea, dysphoria, and other novel subjective negative experiences
Serious Adverse Events | Time of initial intranasal drug administration to 2 hours post intranasal drug administration
  Serious adverse events include: apnea, assisted ventilation, bradypnea, cyanosis, dissociation, emergence reaction, hypotension, laryngospasm, myoclonus, seizure, and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Nshom, MD, Study Director — Cameroon Baptist Convention Health; Michael Runyon, MD, Study Chair — Carolinas Medical Center; James R Young, MD, Principal Investigator — Carolinas Medical Center; Stacy Reynolds, MD, Study Director — Carolinas Medical Center; Hendry R Sawe, MD, Study Director — Muhimbili University of Health and Allied Sciences; Juma Mfinanga, MD, Study Director — Mihumbili National Hospital
Locations (2):
- Mbingo Baptist Hospital, Bamenda, Northwest Province, Cameroon
- Muhimbili National Hospital, Dar es Salaam, Tanzania

REFERENCES:
- [Background] Alli NA, Patel M, Alli HD, Bassa F, Coetzee MJ, Davidson A, Essop MR, Lakha A, Louw VJ, Novitzky N, Philip V, Poole JE, Wainwright RD. Recommendations for the management of sickle cell disease in South Africa. S Afr Med J. 2014 Nov;104(11):743-51. doi: 10.7196/samj.8470. PMID 25909112
- [Background] Diallo D, Tchernia G. Sickle cell disease in Africa. Curr Opin Hematol. 2002 Mar;9(2):111-6. doi: 10.1097/00062752-200203000-00005. PMID 11844993
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Gill FM, Sleeper LA, Weiner SJ, Brown AK, Bellevue R, Grover R, Pegelow CH, Vichinsky E. Clinical events in the first decade in a cohort of infants with sickle cell disease. Cooperative Study of Sickle Cell Disease. Blood. 1995 Jul 15;86(2):776-83. PMID 7606007
- [Background] Olabode JO, Shokunbi WA. Types of crises in sickle cell disease patients presenting at the haematology day care unit (HDCU), University College Hospital (UCH), Ibadan. West Afr J Med. 2006 Oct-Dec;25(4):284-8. PMID 17402517
- [Background] Quinn CT, Shull EP, Ahmad N, Lee NJ, Rogers ZR, Buchanan GR. Prognostic significance of early vaso-occlusive complications in children with sickle cell anemia. Blood. 2007 Jan 1;109(1):40-5. doi: 10.1182/blood-2006-02-005082. Epub 2006 Aug 29. PMID 16940426
- [Background] Ogun GO, Ebili H, Kotila TR. Autopsy findings and pattern of mortality in Nigerian sickle cell disease patients. Pan Afr Med J. 2014 May 8;18:30. doi: 10.11604/pamj.2014.18.30.4043. eCollection 2014. PMID 25368719
- [Background] Makani J, Ofori-Acquah SF, Nnodu O, Wonkam A, Ohene-Frempong K. Sickle cell disease: new opportunities and challenges in Africa. ScientificWorldJournal. 2013;2013:193252. doi: 10.1155/2013/193252. Epub 2013 Sep 19. PMID 25143960
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Background] Kohrs R, Durieux ME. Ketamine: teaching an old drug new tricks. Anesth Analg. 1998 Nov;87(5):1186-93. doi: 10.1097/00000539-199811000-00039. No abstract available. PMID 9806706
- [Background] Green SM, Clem KJ, Rothrock SG. Ketamine safety profile in the developing world: survey of practitioners. Acad Emerg Med. 1996 Jun;3(6):598-604. PMID 8727631
- [Background] Reich DL, Silvay G. Ketamine: an update on the first twenty-five years of clinical experience. Can J Anaesth. 1989 Mar;36(2):186-97. doi: 10.1007/BF03011442. PMID 2650898
- [Background] White JM, Ryan CF. Pharmacological properties of ketamine. Drug Alcohol Rev. 1996 Jun;15(2):145-55. doi: 10.1080/09595239600185801. PMID 16203365
- [Background] Smith DC, Mader TJ, Smithline HA. Low dose intravenous ketamine as an analgesic: a pilot study using an experimental model of acute pain. Am J Emerg Med. 2001 Oct;19(6):531-2. doi: 10.1053/ajem.2001.27152. No abstract available. PMID 11593484
- [Background] Graudins A, Meek R, Egerton-Warburton D, Oakley E, Seith R. The PICHFORK (Pain in Children Fentanyl or Ketamine) trial: a randomized controlled trial comparing intranasal ketamine and fentanyl for the relief of moderate to severe pain in children with limb injuries. Ann Emerg Med. 2015 Mar;65(3):248-254.e1. doi: 10.1016/j.annemergmed.2014.09.024. Epub 2014 Nov 18. PMID 25447557
- [Background] Fu ES, Miguel R, Scharf JE. Preemptive ketamine decreases postoperative narcotic requirements in patients undergoing abdominal surgery. Anesth Analg. 1997 May;84(5):1086-90. doi: 10.1097/00000539-199705000-00024. PMID 9141936
- [Background] Nesher N, Ekstein MP, Paz Y, Marouani N, Chazan S, Weinbroum AA. Morphine with adjuvant ketamine vs higher dose of morphine alone for immediate postthoracotomy analgesia. Chest. 2009 Jul;136(1):245-252. doi: 10.1378/chest.08-0246. Epub 2008 Aug 27. PMID 18753471
- [Background] Wolfe TR, Braude DA. Intranasal medication delivery for children: a brief review and update. Pediatrics. 2010 Sep;126(3):532-7. doi: 10.1542/peds.2010-0616. Epub 2010 Aug 9. PMID 20696726
- [Background] Pandey RK, Bahetwar SK, Saksena AK, Chandra G. A comparative evaluation of drops versus atomized administration of intranasal ketamine for the procedural sedation of young uncooperative pediatric dental patients: a prospective crossover trial. J Clin Pediatr Dent. 2011 Fall;36(1):79-84. doi: 10.17796/jcpd.36.1.1774746504g28656. PMID 22900449
- [Background] Donnelly RF. Stability of diluted ketamine packaged in glass vials. Can J Hosp Pharm. 2013 May;66(3):198. doi: 10.4212/cjhp.v66i3.1259. No abstract available. PMID 23814289
- [Background] Walker SE, Law S, DeAngelis C. Stability and compatibility of hydromorphone and ketamine in normal saline. Can J Hosp Pharm. 2001;54(3):191-199.
- [Background] Arya R, Gulati S, Kabra M, Sahu JK, Kalra V. Intranasal versus intravenous lorazepam for control of acute seizures in children: a randomized open-label study. Epilepsia. 2011 Apr;52(4):788-93. doi: 10.1111/j.1528-1167.2010.02949.x. Epub 2011 Jan 28. PMID 21275979
- [Background] Borland M, Jacobs I, King B, O'Brien D. A randomized controlled trial comparing intranasal fentanyl to intravenous morphine for managing acute pain in children in the emergency department. Ann Emerg Med. 2007 Mar;49(3):335-40. doi: 10.1016/j.annemergmed.2006.06.016. Epub 2006 Oct 25. PMID 17067720
- [Background] Tayebati SK, Nwankwo IE, Amenta F. Intranasal drug delivery to the central nervous system: present status and future outlook. Curr Pharm Des. 2013;19(3):510-26. PMID 23116337
- [Background] Pires A, Fortuna A, Alves G, Falcao A. Intranasal drug delivery: how, why and what for? J Pharm Pharm Sci. 2009;12(3):288-311. doi: 10.18433/j3nc79. PMID 20067706
- [Background] Green SM, Roback MG, Krauss B, Brown L, McGlone RG, Agrawal D, McKee M, Weiss M, Pitetti RD, Hostetler MA, Wathen JE, Treston G, Garcia Pena BM, Gerber AC, Losek JD; Emergency Department Ketamine Meta-Analysis Study Group. Predictors of airway and respiratory adverse events with ketamine sedation in the emergency department: an individual-patient data meta-analysis of 8,282 children. Ann Emerg Med. 2009 Aug;54(2):158-68.e1-4. doi: 10.1016/j.annemergmed.2008.12.011. Epub 2009 Feb 7. PMID 19201064
- [Background] Yanagihara Y, Ohtani M, Kariya S, Uchino K, Hiraishi T, Ashizawa N, Aoyama T, Yamamura Y, Yamada Y, Iga T. Plasma concentration profiles of ketamine and norketamine after administration of various ketamine preparations to healthy Japanese volunteers. Biopharm Drug Dispos. 2003 Jan;24(1):37-43. doi: 10.1002/bdd.336. PMID 12516077
- [Background] Malinovsky JM, Servin F, Cozian A, Lepage JY, Pinaud M. Ketamine and norketamine plasma concentrations after i.v., nasal and rectal administration in children. Br J Anaesth. 1996 Aug;77(2):203-7. doi: 10.1093/bja/77.2.203. PMID 8881626
- [Background] Tsze DS, Steele DW, Machan JT, Akhlaghi F, Linakis JG. Intranasal ketamine for procedural sedation in pediatric laceration repair: a preliminary report. Pediatr Emerg Care. 2012 Aug;28(8):767-70. doi: 10.1097/PEC.0b013e3182624935. PMID 22858745
- [Background] Herd DW, Anderson BJ, Keene NA, Holford NH. Investigating the pharmacodynamics of ketamine in children. Paediatr Anaesth. 2008 Jan;18(1):36-42. doi: 10.1111/j.1460-9592.2007.02384.x. PMID 18095964
- [Background] Yeaman F, Oakley E, Meek R, Graudins A. Sub-dissociative dose intranasal ketamine for limb injury pain in children in the emergency department: a pilot study. Emerg Med Australas. 2013 Apr;25(2):161-7. doi: 10.1111/1742-6723.12059. Epub 2013 Mar 20. PMID 23560967
- [Background] Johansson J, Sjoberg J, Nordgren M, Sandstrom E, Sjoberg F, Zetterstrom H. Prehospital analgesia using nasal administration of S-ketamine--a case series. Scand J Trauma Resusc Emerg Med. 2013 May 14;21:38. doi: 10.1186/1757-7241-21-38. PMID 23672762
- [Background] Ambe JP, Mava Y, Chama R, Farouq G, Machoko Y. Clinical features of sickle cell anaemia in northern nigerian children. West Afr J Med. 2012 Apr-Jun;31(2):81-5. PMID 23208475
- [Background] Piel FB, Hay SI, Gupta S, Weatherall DJ, Williams TN. Global burden of sickle cell anaemia in children under five, 2010-2050: modelling based on demographics, excess mortality, and interventions. PLoS Med. 2013;10(7):e1001484. doi: 10.1371/journal.pmed.1001484. Epub 2013 Jul 16. PMID 23874164
- [Background] Aloni MN, Nkee L. Challenge of managing sickle cell disease in a pediatric population living in kinshasa, democratic republic of congo: a sickle cell center experience. Hemoglobin. 2014;38(3):196-200. doi: 10.3109/03630269.2014.896810. Epub 2014 Mar 26. PMID 24669956
- [Background] Govoni MM. Mandatory education and credentialing for dental assistants: is it the answer to the manpower crisis? Dent Assist (1931). 1990 Jul-Aug;59(4):9-12. PMID 2209936
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Background] Nielsen BN, Friis SM, Romsing J, Schmiegelow K, Anderson BJ, Ferreiros N, Labocha S, Henneberg SW. Intranasal sufentanil/ketamine analgesia in children. Paediatr Anaesth. 2014 Feb;24(2):170-80. doi: 10.1111/pan.12268. Epub 2013 Oct 1. PMID 24118506
- [Background] Palermo TM, Riley CA, Mitchell BA. Daily functioning and quality of life in children with sickle cell disease pain: relationship with family and neighborhood socioeconomic distress. J Pain. 2008 Sep;9(9):833-40. doi: 10.1016/j.jpain.2008.04.002. Epub 2008 Jun 12. PMID 18550443
- [Background] PedsQL Sickle Cell Disease Module, Version 3.0. 1998 JW Varni, Ph.D. (http://www.proqolid.org/instruments/pediatric_quality_of_life_inventory_sickle_cell_disease_module_pedsql_sickle_cell_disease_module)
- [Background] Chien YW, Su KSE, Chang SF, Chapter 1: Anatomy and Physiology of the Nose. Nasal Systemic Drug Delivery, 1989. Dekker, New York: p. 1-26.
- [Background] Who.int,. "WHO | WHO Model Lists Of Essential Medicines." N.p., 2015. Web. 20 July 2015.
- [Background] American Pain Society (1999a) Guideline for the Management of Acute and Chronic Pain in Sickle Cell Disease. American Pain Society, Glenview, IL.
- [Background] World Health Organisation, "Sickle cell anaemia. Agenda item 11.4," in 59th World Health Assembly, 27 May 2006, World Health Organisation, Geneva, Switzerland, 2006.
- [Derived] Young JR, Sawe HR, Mfinanga JA, Nshom E, Helm E, Moore CG, Runyon MS, Reynolds SL. Subdissociative intranasal ketamine plus standard pain therapy versus standard pain therapy in the treatment of paediatric sickle cell disease vaso-occlusive crises in resource-limited settings: study protocol for a randomised controlled trial. BMJ Open. 2017 Jul 10;7(7):e017190. doi: 10.1136/bmjopen-2017-017190. PMID 28698351